CLINICAL TRIAL: NCT01367262
Title: Disposition of [14C]-LY2886721 Following Oral Administration in Healthy Human Subjects
Brief Title: Disposition of Carbon-14-Labeled LY2886721 ([^14C]-LY2886721) Following Oral Administration in Healthy Human Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 13736; I4O-MC-BACD (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-06-03; First posted 2011-06-07 (Estimated); Results first posted 2019-09-13 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-05

CONDITIONS: Healthy Volunteers
Keywords: Absorption; Distribution; Metabolism; Excretion
MeSH Terms: interventions — N-(3-(2-amino-4a,5,7,7a-tetrahydro-4H-furo(3,4-d)(1,3)thiazin-7a-yl)-4-fluorophenyl)-5-fluoropicolinamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiolabeled LY2886721 (Experimental): Single 25 milligram (mg) oral dose containing 80 microCuries of radiolabeled LY2886721
  Interventions: Drug: LY2886721

INTERVENTIONS:
Drug: LY2886721 — Administered orally

SUMMARY:
This open-label study is being conducted to determine the metabolism and physiological disposition of radiolabeled LY2886721 after a single dose in healthy male participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males as determined by medical history and physical examination
* Males will be sterile (including vasectomy) or if the participant is not sterile and is sexually active, he will agree to use from check-in until 3 months after exit/discharge, 1 of the following approved methods of contraception: a male condom with spermicide, a sterile sexual partner, use by female sexual partner of an intrauterine device with spermicide, a female condom with spermicide, contraceptive sponge with spermicide, a diaphragm with spermicide, a cervical cap with spermicide, or oral, implantable, transdermal, intravaginal, or injectable contraceptives
* Have a body mass index of 19 to 30 kilograms per square meter (kg/m^2)
* Have clinical laboratory test results within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator
* Have venous access sufficient to allow for blood sampling
* Have normal blood pressure and heart rate (sitting)
* Experience a minimum of at least 1 bowel movement per day
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures
* Have given written informed consent approved by Lilly and the institutional review board (IRB) governing the site

Exclusion Criteria:

* Are currently enrolled in, have completed, or discontinued within the last 30 days from, a clinical trial involving an investigational product other than the investigational product used in this study; or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have known allergies to LY2886721, related compounds, or any components of the formulation
* Are persons who have previously received the investigational product in this study, have completed or withdrawn from this study or any other study investigating LY2886721
* Have a Bazett's corrected QT (QTcB) interval value of >450 milliseconds (msec) or any abnormality in the 12-lead electrocardiogram (ECG) increases the risks associated with participating in the study
* Have an abnormal blood pressure
* Have a history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* Show evidence of human immunodeficiency virus (HIV) infection and/or positive HIV antibodies
* Show evidence of hepatitis C and/or positive hepatitis C antibody
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen
* Intend to use prescription medication, over-the-counter medication, or herbal preparations containing St. John's Wort, kava, garlic, ginger, ginko biloba, or guarana within 14 days prior to admission
* Eating of grapefruit or grapefruit-containing foods, or drinking grapefruit-containing juices within 7 days prior to dosing or any time during the study
* Have used any tobacco- or nicotine-containing products (including, but not limited to, cigarettes, pipes, cigars, chewing tobacco, nicotine patches, nicotine lozenges, or nicotine gum) within 6 months prior to dosing
* Have donated blood of more than 500 milliliters (mL) within the last month
* Have an average weekly alcohol intake that exceeds 21 units per week (males up to age 65), or are unwilling to stop alcohol consumption from 48 hours prior to check-in until end of study [1 unit = 12 ounces (oz) or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits]
* Show evidence of significant active neuropsychiatric disease, in particular evidence of significant medical or psychiatric illness within the past 12 months. Have any other condition that would preclude participation in the study
* Have a history or presence of epilepsy, a history of seizures, any known brain abnormalities, and a history of significant brain injury
* Have participated in a [^14C] study within the last 6 months prior to check-in for this study. The total exposure from this study and the previous study must be within the Code of Federal Regulations (CFR) recommended levels considered safe (per 21 CFR 361.1), less than 5,000 millirems (mrem)/year whole body annual exposure
* Exposure to significant radiation within 12 months prior to dose (for example, serial X-ray or computed tomography scans, barium meal, current employment in a job requiring radiation exposure monitoring)
* Have a history of clinically significant adverse drug reactions or "drug allergy" to more than 3 types of systemically administered medications (all penicillins and cephalosporins may be considered 1 type of medication for this purpose)
* Have a history of, or current, significant ophthalmological disease
* Have evidence of active renal disease (for example, diabetic renal disease, polycystic kidney disease) or creatinine clearance of <80 milliliters per minute (mL/min) as calculated by Cockcroft-Gault equation: Men: (140-age)*weight in kilograms (kg)/72*[serum creatinine in milligrams per deciliter (mg/dL)]

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2011-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 am - 5 pm Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were considered to have completed the study at 9 days postdose or earlier if ≥90% of administered radioactivity recovered or 24-hour urine and fecal samples from 2 consecutive collections each had radioactivity levels <1.0% of total administered radioactivity in urine and feces combined.
Groups:
- [^14C]-LY2886721: Single 25-milligram (mg) LY2886721 dose containing approximately 80 microCuries (μCi) of carbon-14-labeled LY2886721 ([^14C]-LY2886721), administered as an oral solution.
Period: Overall Study
Arm/Group | [^14C]-LY2886721
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- [^14C]-LY2886721: Single 25-mg LY2886721 dose containing approximately 80 μCi of [^14C]-LY2886721, administered as an oral solution.
Arm/Group | [^14C]-LY2886721
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.2 (12.4)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Males | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Urinary and Fecal Excretion of LY2886721 Radioactivity Over Time
Description: Urinary and fecal excretion of LY2886721 radioactivity over time was expressed as a percentage of the total radioactive dose administered. The amount of drug-related material excreted in urine and feces (Ae) at a specific collection interval (i) was calculated as the product of radioactivity concentration and volume or weight. The Ae values for each collection interval were then summed and calculated as Total Ae=Ae(i1)+Ae(i2)+Ae(in). The percentage of the total radiolabeled dose administered that was excreted in feces or urine=[(Total Ae)/(Total radioactive dose administered)]*100.
Time Frame: Predose up to 7 days (168 hours) postdose
Population: All enrolled participants.
Measure: Mean (Standard Deviation); unit: percentage of radioactive dose
Arm/Group | [^14C]-LY2886721
Number analyzed (Participants) | 6
percentage of radioactive dose
  Urine | 85.7 (2.44)
  Feces | 8.86 (0.868)

2. Secondary Outcome: Plasma Pharmacokinetics (PK) of LY2886721: Area Under the Concentration-Time Curve From Time 0 to Infinity [AUC(0 to Inf)]
Time Frame: Predose up to 4 days (96 hours) postdose
Population: All enrolled participants.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanograms per milliliter (h*ng/mL)
Arm/Group | [^14C]-LY2886721
Number analyzed (Participants) | 6
hours*nanograms per milliliter (h*ng/mL) | 681 (13)

3. Secondary Outcome: PK of Radioactivity: AUC(0 to Inf)
Description: AUC(0 to inf) for plasma and whole blood total radioactivity is reported as hours*nanogram equivalents per milliliter (h*ng Eq/mL).
Time Frame: Predose up to 4 days (96 hours) postdose
Population: All enrolled participants.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng Eq/mL
Arm/Group | [^14C]-LY2886721
Number analyzed (Participants) | 6
h*ng Eq/mL
  Plasma Total Radioactivity | 3310 (13)
  Whole Blood Total Radioactivity | 2470 (13)

4. Secondary Outcome: Plasma PK of LY2886721: Maximum Observed Concentration (Cmax)
Time Frame: Predose up to 4 days (96 hours) postdose
Population: All enrolled participants.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | [^14C]-LY2886721
Number analyzed (Participants) | 6
nanograms per milliliter (ng/mL) | 56.3 (15)

5. Secondary Outcome: PK of Radioactivity: Cmax
Description: The Cmax of total radioactivity in plasma and whole blood are reported as nanogram equivalents per milliliter (ng Eq/mL).
Time Frame: Predose up to 4 days (96 hours) postdose
Population: All enrolled participants.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng Eq/mL
Arm/Group | [^14C]-LY2886721
Number analyzed (Participants) | 6
ng Eq/mL
  Plasma Total Radioactivity | 218 (15)
  Whole Blood Total Radioactivity | 165 (16)

6. Secondary Outcome: Relative Abundance of LY2886721 and the Metabolites of LY2886721 in Plasma
Description: The metabolites of LY2886721 were identified using a high performance liquid chromatography (HPLC) chromatogram. The relative abundance of LY2886721 and its metabolites in plasma were reported as a percentage of recovered radioactivity and calculated by dividing the sum of the radioactive content of fractions contributing to a particular peak by the sum of the radioactive content of all fractions in the radio chromatogram, then multiplying by 100. Radioactivity corresponds to 80 μCi [^14C]-LY2886721.
Time Frame: 1 to 8 hours postdose
Population: All enrolled participants.
Measure: Mean (Standard Deviation); unit: percentage of recovered radioactivity
Arm/Group | [^14C]-LY2886721
Number analyzed (Participants) | 6
percentage of recovered radioactivity
  LY2886721 (parent) 1-hour(h) Postdose | 42.1 (9.8)
  Predominant Metabolite 1h Postdose | 18.0 (6.6)
  LY2886721 (parent) 2h Postdose | 38.3 (6.4)
  Predominant Metabolite 2h Postdose | 15.7 (6.5)
  LY2886721 (parent) 4h Postdose | 37.2 (6.6)
  Predominant Metabolite 4h Postdose | 13.7 (3.1)
  LY2886721 (parent) 8h Postdose | 39.4 (12.9)
  Predominant Metabolite 8h Postdose | 15.2 (2.8)

7. Secondary Outcome: Relative Abundance of LY2886721 and the Metabolites of LY2886721 in Urine
Description: The metabolites of LY2886721 were identified using an HPLC chromatogram. The relative abundance of LY2886721 and its metabolites in urine were reported as a percentage of recovered radioactivity and calculated by dividing the sum of the radioactive content of fractions contributing to a particular peak by the sum of the radioactive content of all fractions in the radio chromatogram, then multiplying by 100. Radioactivity corresponds to 80 μCi [^14C]-LY2886721.
Time Frame: 0 to 72 hours postdose
Population: All enrolled participants.
Measure: Mean (Standard Deviation); unit: percentage of recovered radioactivity
Arm/Group | [^14C]-LY2886721
Number analyzed (Participants) | 6
percentage of recovered radioactivity
  LY2886721 (parent) | 12.3 (3.7)
  Predominant Metabolite | 36.4 (3.6)

8. Secondary Outcome: Relative Abundance of LY2886721 and the Metabolites of LY2886721 in Feces
Description: The metabolites of LY2886721 were identified using an HPLC chromatogram. The relative abundance of LY2886721 and its metabolites in feces were reported as a percentage of recovered radioactivity and calculated by dividing the sum of the radioactive content of fractions contributing to a particular peak by the sum of the radioactive content of all fractions in the radio chromatogram, then multiplying by 100. Radioactivity corresponds to 80 μCi [^14C]-LY2886721.
Time Frame: 0 to 144 hours postdose
Population: All enrolled participants.
Measure: Mean (Standard Deviation); unit: percentage of recovered radioactivity
Arm/Group | [^14C]-LY2886721
Number analyzed (Participants) | 6
percentage of recovered radioactivity
  LY2886721 (parent) | NA (NA) — The relative abundance of LY2886721 in feces was not determined because LY2886721 was below the limit of quantitation.
  Metabolites | 4.1 (2.4)

ADVERSE EVENTS:
Arm/Group | [^14C]-LY2886721
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 3/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | [^14C]-LY2886721 (N=6)
Application site erythema (General disorders) | 2 (2)
Vessel puncture site haematoma (General disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (2)

LIMITATIONS AND CAVEATS:
Assay sensitivity of plasma and whole blood radioactivity were not generally quantifiable after 24-hours postdose. Consequently, the AUC(0-inf) estimate for total radioactivity in plasma and whole blood should be considered underestimated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days